CLINICAL TRIAL: NCT04940572
Title: AUDIOWOLF: A Phase II, Open-label, Efficacy Study of Daily Administration of Sodium Valproate in Patients Clinically Affected by Wolfram Syndrome Due to Monogenic Mutation.
Brief Title: Efficacy Study of Daily Administration of VPA in Patients Affected by Wolfram Syndrome
Acronym: AUDIOWOLF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Etude des Cellules Souches (Other)
Collaborators: Genethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004594-43
Record Dates: First submitted 2021-05-11; First posted 2021-06-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Wolfram Syndrome
MeSH Terms: conditions — Wolfram Syndrome | interventions — Valproic Acid

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depakine (VPA) (Experimental): Depakine Chrono 500 mg (VPA)
  VPA will be administered orally:
  * From D1 to D3: During the first week 10-15 mg sodium valproate/kg bodyweight per day will be taken daily.
  * From D3 to W156: The dose will be increased every 3 days in steps of 10 mg sodium valproate/kg bodyweight per day with VPA plasma concentration monitoring until the total daily dose corresponding to the optimal plasma level between 40 and 100 mg/l (ie, 300 to 700 micromol/l) is reached, till the 156 weeks corresponding to the end of treatment (EOT) visit.
  The total daily dose will be taken in one or two doses during meals.
  Interventions: Drug: Depakine

INTERVENTIONS:
Drug: Depakine — Refer to arm description.

SUMMARY:
Open label, phase II study non randomized single group assignment of 20 evaluable patients 13 years and older, over 37,5 kg body-weight, with sensorineural hearing loss of at least 20 dB at 8 kHz in high frequency average (HFA), and with documented genetic mutations in the WFS1 gene and with at least one other major documented clinical symptom pertaining to Wolfram syndrome (i.e. diabetes mellitus, diabetes insipidus, optic atrophy). Every patients will receive over three years a treatment by VPA (Depakine chrono).

DETAILED DESCRIPTION:
Open label, phase II study non randomized single group assignment of 20 evaluable patients 13 years and older, over 37,5 kg body-weight, with sensorineural hearing loss of at least 20 dB at 8 kHz in high frequency average (HFA), AND with documented genetic mutations in the WFS1 gene AND with at least one other major documented clinical symptom pertaining to Wolfram syndrome (i.e. diabetes mellitus, diabetes insipidus, optic atrophy). Every patients will receive over three years a treatment by VPA (Depakine chrono).

The effective dose and duration of this 3 years therapy has to be determined individually with the aim to obtain preservation of auditory function defined as no decrease higher than 5 dB on one ear compared to baseline at 8 kHz on high frequencies average and to reduce the dose of insulin and/or desmopressin needed, therefore monitoring of the patients plasma concentration of VPAis required for dose adjustment.

Generally a plasma level between 40 and 100 mg/l (ie, 300 to 700 micromol/l) sodium valproate is aimed to be reached.

Initially 10-15 mg of sodium valproate/kg bodyweight per day will be taken in one or two doses during meals. The dose will then be increased every 3 days in steps of 10 mg sodium valproate/kg bodyweight per day till the optimal plasma level is reached but does not exceed 100 milligrams per liter (ie, 700 micromol/l) during 156 weeks (refer to Appendix 5).

Analysis will compare Pure tone audiometry (PTA), Speech interference index (SII) and High frequency pure tone audiometry hearing test between baseline and final visit.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a definite diagnosis of Wolfram syndrome, as determined by the following:

   * Documented diabetes mellitus diagnosed under 16 completed years according to WHO or ADA criteria OR documented optic atrophy diagnosed under 16 completed years AND Documented functionally relevant mutations on one or both alleles of the WFS1 gene based on historical test results (if available) or from a qualified laboratory at screening
2. The patient has sensorineural hearing loss of at least 20 db at 8 kHz in HFA
3. The patient is 13 years of age or older, and has a body-weight over 37.5 kg
4. Written informed consent for the principal study
5. Women of childbearing potential who are prescribed with sodium valproate must use effective contraception without interruption during the entire duration of treatment and at least 90 days after last administration . These patients will be provided with comprehensive information on pregnancy prevention and will be referred for contraceptive advice if they are not using effective contraception. At least one effective method of contraception (preferably a user independent form such as an intra-uterine device or implant) or two complementary forms of contraception including a barrier method should be used.
6. Women with childbearing potential are required to have a confirmed negative blood pregnancy test before starting medication administration at baseline. Women with childbearing potential agree to repeat blood pregnancy tests during at each study visit.
7. Sexually active men with a female partner of childbearing potential must agree to the use of condoms and the use of a effective method of contraception by the female partner.
8. Patient willing and able to meet all protocol defined visits for the duration of the Trial.
9. Patients with active hearing implants, containing a magnetic system are allowed to participate to study, and will not have MRI during study participation.

Exclusion Criteria:

1. The patient is unable or unwilling to comply with the protocol requirements
2. The patient has received treatment with any investigational drug within the 30 days prior to the screening visit
3. The patient is currently taking VPA
4. The patient has an history of allergy or hypersensitivity to VPA or its excipients/ingredients
5. The patient is known to be affected by a pathology for which the symptoms or associated treatments can alter the hearing function and/or affect the ear
6. The patient has clinically significant non-Wolfram related CNS involvement which is judged by the Investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments
7. The patient has a contra-indication to VPA: mitochondrial disorders caused by mutations in the nuclear gene encoding the mitochondrial enzyme polymerase γ (POLG), e.g. Alpers-Huttenlocher Syndrome, active liver disease, personal or family history of liver dysfunction related to known genetic disorders, porphyria, lactose intolerance, the Lapp lactase deficiency, glucose- galactose malabsorption, urea cycle disorders…
8. Any other acute or chronic medical, psychiatric, social situation or laboratory result that, based on Investigator's judgment, would jeopardize patient safety during trial participation, cause inability to comply with the protocol, or affect the Trial participation
9. The patient has a known history of central apnea
10. An unwillingness on the part of male patients to use highly effective form of birth control if engaging in sexual intercourse with a woman who could become pregnant from the time of the first dose of study medication until completion of follow-up procedures.
11. An unwillingness on the part of female patients to use highly effective form of birth control if engaging in sexual intercourse and to have frequent pregnancy tests during treatment and until completion of follow-up procedures.
12. The patient is currently pregnant or breastfeeding
13. The patient is swallowing disorders

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Preservation of auditory function. | Baseline - Week 156
  Preservation of auditory function defined as no decrease higher than 5 dB in hearing at 8 kHz in high frequency average (HFA) over three years in patients with Wolfram syndrome with a deficit of at least 20d dB at 8 kHz treated with VPA at optimal dose corresponding to the plasma level between 40 and 100 mg/l (ie, 300 to 700 micro mol/l).

SECONDARY OUTCOMES:
Safety endpoint | Baseline - Week 156
  Overall incidence of adverse events and serious adverse events as well as laboratory assessments will be evaluated for each group and for the study as a whole.
Ventral Pons Volume measure | Baseline - Week 156
  Ventral Pons Volume measured and recorded in mm3 by standardised analysis of MRI at baseline, at visit 8 (Week 52) and at the final visit.
Insulin and or desmopressin requirements | Baseline - Week 156
  Insulin and or desmopressin requirements will be assessed whenever the patient is under one or both treatments in order to document potential benefit from VPA on diabetes mellitus or diabetes insipidus
Visual acuity assessment | Baseline - Week 156
  Visual acuity will be assessed using standard ETDRS measures and visual field recording at baseline, every six months during the first year of follow-up and at the final visit
Retinal nerve thikness measure | Baseline - Week 156
  Retinal nerve thikness measured by OCT measures at baseline, every six months during the first year of follow-up and at the final visit
Balance measured by Mini-BESTest | Baseline - Week 156
  Balance, measured by Mini-BESTest (Appendix 1) at baseline, at visit 8 (Week 52) and at the final visit.
Quality of sleep assessment on pediatric population - Qualitative questionnaire (no scale) | Baseline - Week 156
  Sleep will be investigated by Pediatric Sleep Questionnaire at baseline, at visit 8 (Week 52) and at final visit.
Quality of sleep assessment on adult population - Qualitative questionnaire (no scale) | Baseline - Week 156
  Sleep will be investigated by Pittsburg Sleep Quality Index Self-Report on adult population at baseline, at visit 8 (Week 52) and at final visit.

CONTACTS AND LOCATIONS:
Locations (2):
- HEGP, Paris, France
- Centro periférico de Especialidades de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No